CLINICAL TRIAL: NCT02937857
Title: A Multicenter, Randomized, Open Label, Add-on Study to Assess Efficacy and Safety of Xiyanping Injection in Subjects With Pediatric Bronchitis
Brief Title: An Add-on Study to Evaluate the Efficacy and Safety of Xiyanping Injection in Pediatric Bronchitis Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JXQF-XYP-1606
Record Dates: First submitted 2016-09-20; First posted 2016-10-19 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2016-09

CONDITIONS: Bronchitis
MeSH Terms: conditions — Bronchitis | interventions — Anti-Asthmatic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment only (Active Comparator): Standard treatment only such as antiasthmatic, expectorant and antipyretic
  Interventions: Drug: Standard treatment only
- Standard treatment+Xiyanping injection (Experimental): Standard Treatment such as antiasthmatic, expectorant and antipyretic plus Xiyanping injection intravenous administration of 0.2-0.4mL/kg/day ,QD for 5 days.
  Interventions: Drug: Standard treatment+Xiyanping injection

INTERVENTIONS:
Drug: Standard treatment only — standard treatment， such as antiasthmatic,expectorant,antipyretic
  Other Names: antiasthmatic,expectorant,antipyretic
  Arms: Standard treatment only
Drug: Standard treatment+Xiyanping injection — standard treatment+Xiyanping injection:standard treatment， such as antiasthmatic, expectorant and antipyretic plus Xiyanping injection,0.2-0.4mL/kg/day,qd for 5 days.
  Other Names: antiasthmatic,expectorant,antipyretic + Xiyanping injection
  Arms: Standard treatment+Xiyanping injection

SUMMARY:
This is a multicenter, randomized, open Label,add-on study.

DETAILED DESCRIPTION:
This is an add-on study of efficacy and safety of intravenous injection of Xiyanping injection in subjects with pediatric bronchitis.

The purpose to determine the efficacy and safety of conventional treatment combined with or without Xiyanping injection in the treatment of pediatric bronchitis and to further evaluate the clinical value of Xiyanping injection in shortening the course of pediatric bronchitis

The study will enroll 240 Pediatric bronchitis volunteers, who will be randomized into 2 groups (1:1 ratio): volunteers from the first group will receive Routine treatment for pediatric bronchitis and Xiyanping injection; volunteers from the second group will receive Routine treatment for pediatric bronchitis. Xiyanping injection will be administration as intravenous injection of 0.2-0.4mL/kg/day once daily for 5 days concomitantly with Routine treatment for pediatric bronchitis

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pediatric bronchitis with hospital treatment needed
* Males and female subjects
* Age between 1 and 3 years old
* With fever, cough, gasp and expectoration symptoms
* Have wheeze and/ or mid-fine rales on one's lungs
* White blood cell count < 12 x 109 / L, categorized priority to leukocyte
* C-reactive protein≤8mg/L or normal Super C- reactive protein
* Had experienced ≤48 h course before enrollment
* Previous Wheezing episodes≤2
* Written informed consent

Exclusion Criteria:

* Participants with severe clinical symptoms, meet any of the following：

  * SaO2≤0.92;（2）Shock or disturbance of consciousness;（3） Significantly speed up breathing , rapid pulse accompany with severe respiratory distress; or（4）Repeated occurrence of apnea or slow and irregular respiration;
* Acute infectious disease such as measles, pertussis and influenza
* Participants with bronchial asthma, bronchopneumonia and other respiratory diseases
* Chronic lung diseases
* Participants with complicated pyopneumothorax, airway obstruction, toxic encephalopathy, cardiac failure or respiratory failure
* Participants with complicated severe underlying myocardial, liver, kidney, digestive and hematopoietic system diseases
* Severe malnutrition and history of immune deficiency which may seriously affect the self-limiting process of the course
* Participants with epilepsy and other disturbances of central nervous system
* Participants with congenital diseases and psychosis
* use of any other antiviral drugs within the 2 weeks before enrollment
* use of systemic hormone within the 2 weeks before enrollment
* Participants had a history of allergic constitution and drug allergy; Allergenic to XiYanPing injection and Andrographolide
* Participants participated in other clinical research in the last three months
* Any condition which would make the subject, in the opinion of the investigator or designee, not suitable for the study for any reason

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
time to total score of the clinical symptoms/signs decreased more than 70% from baseline | up to 30 days after the last Administration

SECONDARY OUTCOMES:
The total efficiency rate | Day 3 and Day 5
Time to defervescence | up to 30 days after the last Administration
Day(s) of Hospital Stay | up to 30 days after the last Administration
Signs and Symptoms Score from baseline | up to 30 days after the last Administration
Antibiotic consumption | up to 30 days after the last Administration
  check and record the usage of antibiotic,including durg Utilization Rate and the duration of usage
Usage of Inhaled corticosteroids | up to 30 days after the last Administration
  check and record the usage of Inhaled corticosteroids,including durg Utilization Rate and the duration of usage
Incidence of complication | up to 30 days after the last Administration
  record the incidence of new complication after treatment.
Sputum status | up to 30 days after the last Administration
  record the incidence of expectoration and the day of expectoration disappear
Expenditure of therapeutic drug | up to 30 days after the last Administration
The total expenditure of treatment | up to 30 days after the last Administration
  Expenditure of treatment include the cost of durg, hospitalization,examination
incidence of adverse events | up to 30 days after the last Administration

CONTACTS AND LOCATIONS:
Overall Officials: Liu Han Min, professor, Principal Investigator — Sichuan University
Locations (1):
- Guangzhou women and children health care center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided